CLINICAL TRIAL: NCT00283569
Title: Genetic Epidemiology of Adult-Onset Glioma
Brief Title: Genetic Epidemiology of Adult Onset Glioma
Status: Completed | Type: Observational
Sponsor: Kentuckiana Cancer Institute (Other)
Collaborators: DR. Kathleen Egan (Unknown)
Responsible Party: Renato V. LaRocca, MD, Kentuckiana Cancer Institute
Other Study IDs: mrbt1-03-132; MRBTC2003-01
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Adult-Onset Glioma
Keywords: Glioma
MeSH Terms: conditions — Glioma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, Toe Nail Clippings

INTERVENTIONS:
Other: Mouth Swab, Toe Nail Clippings, Questionnaires — The objective of this study is to establish a clinic based case control study for examination of potential risk factors for primary adult brain tumors.

SUMMARY:
To establish a clinic based case control study for examination of potential risk factors for primary adult brain tumors.

DETAILED DESCRIPTION:
Genetic epidemiology of adult glioma to establish potential risk factors for primary adult brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* primary glioma of any stage
* diagnosed within 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Glioma and a Control
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato V. LaRocca, MD, Principal Investigator — Director
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States